CLINICAL TRIAL: NCT00090103
Title: A Randomized, Double-blind, Parallel Group Study to Investigate the Efficacy and Safety of Treatment With Dutasteride (0.5mg) and Tamsulosin (0.4mg), Administered Once Daily for 4 Years, Alone and Combination, on the Improvement of Symptoms and Clinical Outcome in Men With Moderate to Severe Symptomatic Benign Prostatic Hyperplasia
Brief Title: Benign Prostatic Hyperplasia Trial With Dutasteride And Tamsulosin Combination Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARI40005
Record Dates: First submitted 2004-08-24; First posted 2004-08-26 (Estimated); Results first posted 2010-03-16 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Prostatic Hyperplasia
Keywords: Combination Therapy; dutasteride; BPH
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- dutasteride (Active Comparator): dutasteride 0.5mg once daily
  Interventions: Drug: dutasteride 0.5mg once daily for 4 years
- Combo (Experimental): Combination of dutasteride (0.5mg) and tamsulosin (0.4mg), once daily
  Interventions: Drug: dutasteride 0.5mg once daily for 4 years; Drug: tamsulosin 0.4mg once daily for 4 years
- tamsulosin (Active Comparator): tamsulosin 0.4mg once daily
  Interventions: Drug: tamsulosin 0.4mg once daily for 4 years

INTERVENTIONS:
Drug: dutasteride 0.5mg once daily for 4 years — combination or single agent
  Arms: Combo; dutasteride
Drug: tamsulosin 0.4mg once daily for 4 years — combination agent or single agent
  Other Names: dutasteride; tamsulosin
  Arms: Combo; tamsulosin

SUMMARY:
This study will investigate the efficacy and safety of treatment with dutasteride and tamsulosin, administered once daily for 4 years, alone and in combination, on the improvement of symptoms and clinical outcome in men with moderate to severe symptomatic Benign Prostatic Hyperplasia (BPH). Study visits are every 3 months for up to 4 years (18 clinic visits). Transrectal ultrasound (TRUS) is done annually.

DETAILED DESCRIPTION:
A randomised, double-blind, parallel group study to investigate the efficacy and safety of treatment with Dutasteride (0.5 mg) and Tamsulosin (0.4 mg), administered once daily for 4 years, alone and in combination, on the improvement of symptoms and clinical outcome in men with moderate to severe symptomatic benign prostatic hyperplasia.

ELIGIBILITY:
Inclusion criteria:

* A subject will be considered eligible for inclusion in this study only if all of the following criteria apply:
* males, aged ≥50 years
* clinical diagnosis of BPH by medical history and physical examination, including a digital rectal examination (DRE)
* International Prostate Symptom Score (IPSS) ≥12 points at Screening
* prostate volume ≥30 cc by transrectal ultrasonography; (TRUS)
* total serum Prostate Specific Antigen (PSA) ≥1.5ng/mL at Screening
* maximum flow rate (Qmax) >5 mL/sec and ≤15 mL/sec and minimum voided volume of ≥125 mL at Screening (based on two voids)
* willing and able to give written informed consent and comply with study procedures
* fluent and literate in local language with the ability to read, comprehend and record information on the IPSS, BII and Patient Perception of Study Medication
* able to swallow and retain oral medication
* willing and able to participate in the study for the full 4 years.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* total serum PSA >10.0ng/mL at Screening
* history or evidence of prostate cancer (e.g. positive biopsy or ultrasound, suspicious DRE). Patients with suspicious ultrasound or DRE who have had a negative biopsy within the preceding 6 months and stable PSA are eligible for the study.

Note: If total serum PSA is >4ng/mL and unless PSA value has been stable for at least the past 2 years, the investigator should make every appropriate effort to exclude the possibility of prostate cancer, e.g. further DRE, review TRUS taken within previous month, consider 8-12 core prostate biopsy in accordance with routine clinical practice.

* previous prostatic surgery (including TURP, balloon dilatation, thermotherapy and stent replacement) or other invasive procedures to treat BPH.
* history of flexible/rigid cystoscopy or other instrumentation of the urethra within 7 days prior to the Screening Visit. Routine catheterisation is acceptable with no time restriction.
* history of AUR within 3 months prior to Screening Visit.
* post-void residual volume >250mL (suprapubic ultrasound) at Screening.
* any causes other than BPH, which may in the judgement of the investigator, result in urinary symptoms or changes in flow rate (e.g. neurogenic bladder, bladder neck contracture, urethral stricture, bladder malignancy, acute or chronic prostatitis, or acute or chronic urinary tract infections).
* history of breast cancer or clinical breast examination finding of unclear origin or suggestive of malignancy.
* use of any 5-alpha-reductase inhibitor (e.g. Proscar®, Propecia®, Avodart®), any drugs with antiandrogenic properties (e.g. spironolactone, flutamide, bicalutamide, cimetidine, ketoconazole, metronidazole, progestational agents), or other drugs which affect prostate volume, within past 6 months of the Screening Visit and throughout the study (other than as study medication).
* concurrent use of anabolic steroids
* use of phytotherapy for BPH within 2 weeks of Screening Visit and/or predicted to need phytotherapy during the study.
* use of any alpha-adrenoreceptor blockers (i.e. indoramin, prazosin, terazosin, tamsulosin, alfuzosin and doxazosin) within 2 weeks of Screening Visit and/or predicted to need any alpha blockers other than tamsulosin during the study.

Note: the purpose of this criteria is to be able to standardise baseline symptom severity for all enrolled patients prior to randomisation and not to specifically exclude current alpha-adrenoreceptor blocker users from participation in the study.

* use of any alpha-adrenoreceptor agonists (e.g. pseudoephedrine, phenylephrine, ephedrine) or anticholinergics (e.g. oxybutynin, propantheline) or cholinergics (e.g. bethanecol chloride) within 48 hours prior to all uroflowmetry assessments.
* hypersensitivity to any alpha-/beta- adrenoreceptor blocker or 5-alpha-reductase inhibitor, or other chemically-related drugs.
* concurrent use of drugs known or thought to have an interaction with tamsulosin, e.g. cimetidine and warfarin.
* history of hepatic impairment or abnormal liver function tests at Screening defined as alanine aminotransferase (ALT), aspartate aminotranferase (AST), and/or alkaline phosphatase >2 times the upper limit of normal, or total bilirubin >1.5 times the upper limit of normal (unless associated with predominantly indirect bilirubin elevation or Gilbert's syndrome).
* history of renal insufficiency, or serum creatinine >1.5 times the upper limit of normal or serum creatinine ≥1.5 mg/dL at Screening.
* prior history of malignancies other than basal cell carcinoma or squamous cell carcinoma of the skin within the past 5 years. Subjects with a prior malignancy who have had no evidence of disease for at least the past 5 years are eligible.
* history of any illness that in the opinion of the investigator might confound the results of the study or poses additional risk to the patient.
* any unstable, serious co-existing medical condition(s) including, but not limited to, myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to Screening visit; uncontrolled diabetes or peptic ulcer disease which is uncontrolled by medical management.
* history of postural hypotension, dizziness, vertigo or any other signs and symptoms of orthostasis, which in the opinion of the investigator could be exacerbated by tamsulosin and result in putting the subject at risk of injury.
* history of unsuccessful treatment with tamsulosin or 'first dose' hypotensive episode on initiation of alpha-1-adrenoreceptor antagonist therapy.
* history of unsuccessful treatment with finasteride or dutasteride
* history or current evidence of drug or alcohol abuse within the previous 12 months.
* participation in any investigational or marketed drug trial within 30 days (or 5 half-lives whichever is the longer) preceding the Screening Visit and/or during the course of this study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4844 (Actual)
Dates: Start 2003-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (424):
- United States (101):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Columbiana, Alabama
  - GSK Investigational Site, Hoover, Alabama
  - GSK Investigational Site, Anchorage, Alaska
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Phoenix, Arizona, Arizona
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Concord, California
  - GSK Investigational Site, Glendora, California
  - GSK Investigational Site, Greenbrae, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Laguna Woods, California
  - GSK Investigational Site, Los Angelas, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Modesto, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Bay Pines, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Lake Worth, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, New Smyrna Beach, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orange City, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, Pinecrest, Florida
  - GSK Investigational Site, Saint Augustine, Florida
  - GSK Investigational Site, Spring Hill, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Wellington, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Calhoun, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Belleville, Illinois
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Wheaton, Illinois
  - GSK Investigational Site, Winfield, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Jeffersonville, Indiana
  - GSK Investigational Site, Newburgh, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Murray, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Laurel, Maryland
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Picayune, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Perth Amboy, New Jersey
  - GSK Investigational Site, Somerville, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Bay Shore, New York
  - GSK Investigational Site, Garden City, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Lewiston, New York
  - GSK Investigational Site, Asheboro, North Carolina
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Bismarck, North Dakota
  - GSK Investigational Site, Bellbrook, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Fleetwood, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Athes, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, New Brunfels, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Texarkana, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Bellevue, Washington
  - GSK Investigational Site, Mountlake Terrace, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
- Argentina (3):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad de Buenos Aires
- Belgium (7):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Genk
  - GSK Investigational Site, La Louvière
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Roeselare
- Brazil (4):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Rio de Janeiro, Rio de Janeiro
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, São Paulo, São Paulo
- Bulgaria (3):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (25):
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Saint John, New Brunswick
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Kentville, Nova Scotia
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, Brantford, Ontario
  - GSK Investigational Site, Courtice, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Guelph, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Scarborough Village, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Saint-Jérôme, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Czechia (4):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Roudnice nad Labem
- Denmark (4):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Aarhus N
  - GSK Investigational Site, Fredericia
  - GSK Investigational Site, Randers
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Finland (5):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jakobstad
  - GSK Investigational Site, Kouvola
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Tampere
- France (60):
  - GSK Investigational Site, Bully-les-Mines, Hauts-de-France
  - GSK Investigational Site, Agny
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Annecy
  - GSK Investigational Site, Arras
  - GSK Investigational Site, Athis-Mons
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Bouchemaine
  - GSK Investigational Site, Broglie
  - GSK Investigational Site, Castelneau Le Nez
  - GSK Investigational Site, Chambéry
  - GSK Investigational Site, Chilly-Mazarin
  - GSK Investigational Site, Cournonterral
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Domarin
  - GSK Investigational Site, Épinay-sur-Orge
  - GSK Investigational Site, Évreux
  - GSK Investigational Site, Gif-sur-Yvette
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, La Seyne-sur-Mer
  - GSK Investigational Site, Lamarque
  - GSK Investigational Site, Laval
  - GSK Investigational Site, Le Brusc
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Les Mureaux
  - GSK Investigational Site, Lesparre-Médoc
  - GSK Investigational Site, Linas
  - GSK Investigational Site, Longpont-sur-Orge
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Melun
  - GSK Investigational Site, Meudon
  - GSK Investigational Site, Meylan
  - GSK Investigational Site, Mont-de-Marsan
  - GSK Investigational Site, Montauban
  - GSK Investigational Site, Montpelier
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pontonx Sur Adour
  - GSK Investigational Site, Roanne
  - GSK Investigational Site, Saint-Chamond
  - GSK Investigational Site, Saint-Denis
  - GSK Investigational Site, Saint-Egrève
  - GSK Investigational Site, Saint-Galmier
  - GSK Investigational Site, Saint-Georges-dOrques
  - GSK Investigational Site, Saint-Germain-Lespinasse
  - GSK Investigational Site, Saint-Sébastien-de-Morsent
  - GSK Investigational Site, Sainte-Suzanne
  - GSK Investigational Site, Sanary-sur-Mer
  - GSK Investigational Site, Sarlat-la-Canéda
  - GSK Investigational Site, Seysses
  - GSK Investigational Site, Six-Fours-les-Plages
  - GSK Investigational Site, Suresnes
  - GSK Investigational Site, Toulon
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Vaucresson
  - GSK Investigational Site, Verneuil-sur-Seine
  - GSK Investigational Site, Villejuif
  - GSK Investigational Site, Villeneuve-lès-Maguelone
  - GSK Investigational Site, Vourey
- Germany (44):
  - GSK Investigational Site, Aalen, Baden-Wurttemberg
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Konstanz, Baden-Wurttemberg
  - GSK Investigational Site, Mosbach, Baden-Wurttemberg
  - GSK Investigational Site, Rottweil, Baden-Wurttemberg
  - GSK Investigational Site, Stockach, Baden-Wurttemberg
  - GSK Investigational Site, Aichach, Bavaria
  - GSK Investigational Site, Amberg, Bavaria
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Graefeling, Bavaria
  - GSK Investigational Site, Neu-Ulm, Bavaria
  - GSK Investigational Site, Schongau, Bavaria
  - GSK Investigational Site, Wertingen, Bavaria
  - GSK Investigational Site, Hagenow, Brandenburg
  - GSK Investigational Site, Lauchhammer, Brandenburg
  - GSK Investigational Site, Oranienburg, Brandenburg
  - GSK Investigational Site, Senftenberg, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Alzenau, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Giessen, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Koenigstein, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Schwalbach, Hesse
  - GSK Investigational Site, Delmenhorst, Lower Saxony
  - GSK Investigational Site, Holzminden, Lower Saxony
  - GSK Investigational Site, Oldenburg, Lower Saxony
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Grimmen, Mecklenburg-Vorpommern
  - GSK Investigational Site, Parchim, Mecklenburg-Vorpommern
  - GSK Investigational Site, Dülmen, North Rhine-Westphalia
  - GSK Investigational Site, Stadtlohn, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Hohenstein-Ernsttal, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Hettstedt, Saxony-Anhalt
  - GSK Investigational Site, Merseburg, Saxony-Anhalt
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Apolda, Thuringia
- Greece (4):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Pátrai
  - GSK Investigational Site, Polygyros
  - GSK Investigational Site, Thassaloniki
- Hungary (4):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Sopron
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Veszprém
- GSK Investigational Site, Reykjavik, Iceland
- Israel (5):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Zrifin
- Italy (21):
  - GSK Investigational Site, Catanzaro, Calabria
  - GSK Investigational Site, Avellino, Campania
  - GSK Investigational Site, Castellamare Di Stabia (NA), Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, San Felice A Cancello Caserta, Campania
  - GSK Investigational Site, Torre Del Greco (NA), Campania
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Lecco, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Ivrea (TO), Piedmont
  - GSK Investigational Site, Novara, Piedmont
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Acireale (CT), Sicily
  - GSK Investigational Site, Bagno A Ripoli (FI), Tuscany
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Siena, Tuscany
  - GSK Investigational Site, Portogruaro (VE), Veneto
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Klaipėda
  - GSK Investigational Site, Vilnius
- Mexico (5):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco, Jalisco
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
- Netherlands (17):
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Amstelveen
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Arnhem
  - GSK Investigational Site, Doetinchem
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Etten-Leur
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Hilversum
  - GSK Investigational Site, Hoofddorp
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Tilburg
  - GSK Investigational Site, Veldhoven
  - GSK Investigational Site, Winterswijk
  - GSK Investigational Site, Zwijndrecht
- Norway (9):
  - GSK Investigational Site, Ålesund
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Bodø
  - GSK Investigational Site, Haugesund
  - GSK Investigational Site, Moelv
  - GSK Investigational Site, Nøtterøy
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Porsgrunn
  - GSK Investigational Site, Tønsberg
- Philippines (2):
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
- Poland (4):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Wroclaw
- Portugal (4):
  - GSK Investigational Site, Abrantes
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
  - GSK Investigational Site, S. Martinho Do Bispo
- Puerto Rico (2):
  - GSK Investigational Site, Ponce, Puerto Rico
  - GSK Investigational Site, Santurce, Puerto Rico
- Romania (5):
  - GSK Investigational Site, Arad
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Timișoara
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Rostov-on-Don
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
- Slovakia (6):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
  - GSK Investigational Site, Martin
  - GSK Investigational Site, Skalica
  - GSK Investigational Site, Žilina
- South Africa (4):
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Claremont
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Sunninghill
- South Korea (2):
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- Spain (36):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alava
  - GSK Investigational Site, Alcázar de San Juan (Ciudad Real)
  - GSK Investigational Site, Badajoz
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Ciudad Real
  - GSK Investigational Site, Donostia / San Sebastian
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Gijón
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Jerez de la Frontera
  - GSK Investigational Site, Langreo (Oviedo)
  - GSK Investigational Site, Las Palmas
  - GSK Investigational Site, Las Palmas de Gran Canaria
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Manacor (Palma de Mallorca)
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Mendaro, Guipuzcoa
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Pontevedra
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Santa Cruz de Tenerife
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Tortosa
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vigo (Pontevedra)
  - GSK Investigational Site, Vigo/Pontevedra
  - GSK Investigational Site, Vitoria-Gasteiz
  - GSK Investigational Site, Vizcaya
- Taiwan (5):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- Tunisia (2):
  - GSK Investigational Site, Sousse
  - GSK Investigational Site, Tunis
- Turkey (Türkiye) (3):
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Izmir
  - GSK Investigational Site, Sıhhiye/Ankara
- United Kingdom (11):
  - GSK Investigational Site, Swansea, Glamorgan
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Oxford, Oxfordshire
  - GSK Investigational Site, Chichester, Sussex West
  - GSK Investigational Site, Clydebank, Glasgow
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Edgbaston, Birmingham
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Waterloo, Liverpool
- GSK Investigational Site

REFERENCES:
- [Background] Antonanzas F, Brenes F, Molero JM, Fernandez-Pro A, Huerta A, Palencia R, Cozar JM. [Cost-effectiveness of the combination therapy of dutasteride and tamsulosin in the treatment of benign prostatic hyperlasia in Spain]. Actas Urol Esp. 2011 Feb;35(2):65-71. doi: 10.1016/j.acuro.2010.11.008. Epub 2011 Jan 26. Spanish. PMID 21269736
- [Background] Barkin J, Roehrborn CG, Siami P, Haillot O, Morrill B, Black L, Montorsi F; CombAT Study Group. Effect of dutasteride, tamsulosin and the combination on patient-reported quality of life and treatment satisfaction in men with moderate-to-severe benign prostatic hyperplasia: 2-year data from the CombAT trial. BJU Int. 2009 Apr;103(7):919-26. doi: 10.1111/j.1464-410X.2009.08196.x. Epub 2009 Feb 23. PMID 19239460
- [Background] Bjerklund Johansen TE, Baker TM, Black LK. Cost-effectiveness of combination therapy for treatment of benign prostatic hyperplasia: a model based on the findings of the Combination of Avodart and Tamsulosin trial. BJU Int. 2012 Mar;109(5):731-8. doi: 10.1111/j.1464-410X.2011.10511.x. Epub 2011 Sep 20. PMID 21933326
- [Background] Black L, Grove A, Morrill B. The psychometric validation of a US English satisfaction measure for patients with benign prostatic hyperplasia and lower urinary tract symptoms. Health Qual Life Outcomes. 2009 Jun 19;7:55. doi: 10.1186/1477-7525-7-55. PMID 19545384
- [Background] Chung BH, Roehrborn CG, Siami P, Major-Walker K, Morrill BB, Wilson TH, Montorsi F. Efficacy and safety of dutasteride, tamsulosin and their combination in a subpopulation of the CombAT study: 2-year results in Asian men with moderate-to-severe BPH. Prostate Cancer Prostatic Dis. 2009;12(2):152-9. doi: 10.1038/pcan.2008.49. Epub 2008 Sep 23. PMID 18813219
- [Background] Roehrborn CG, Siami P, Barkin J, Damiao R, Major-Walker K, Nandy I, Morrill BB, Gagnier RP, Montorsi F; CombAT Study Group. The effects of combination therapy with dutasteride and tamsulosin on clinical outcomes in men with symptomatic benign prostatic hyperplasia: 4-year results from the CombAT study. Eur Urol. 2010 Jan;57(1):123-31. doi: 10.1016/j.eururo.2009.09.035. Epub 2009 Sep 19. PMID 19825505
- [Background] Roehrborn CG, Andriole GL, Wilson TH, Castro R, Rittmaster RS. Effect of dutasteride on prostate biopsy rates and the diagnosis of prostate cancer in men with lower urinary tract symptoms and enlarged prostates in the Combination of Avodart and Tamsulosin trial. Eur Urol. 2011 Feb;59(2):244-9. doi: 10.1016/j.eururo.2010.10.040. Epub 2010 Nov 4. PMID 21093145
- [Background] Roehrborn CG, Barkin J, Siami P, Tubaro A, Wilson TH, Morrill BB, Gagnier RP. Clinical outcomes after combined therapy with dutasteride plus tamsulosin or either monotherapy in men with benign prostatic hyperplasia (BPH) by baseline characteristics: 4-year results from the randomized, double-blind Combination of Avodart and Tamsulosin (CombAT) trial. BJU Int. 2011 Mar;107(6):946-54. doi: 10.1111/j.1464-410X.2011.10124.x. Epub 2011 Feb 18. PMID 21332630
- [Background] Roehrborn CG, Wilson TH, Black LK. Quantifying the contribution of symptom improvement to satisfaction of men with moderate to severe benign prostatic hyperplasia: 4-year data from the CombAT trial. J Urol. 2012 May;187(5):1732-8. doi: 10.1016/j.juro.2011.12.083. Epub 2012 Mar 15. PMID 22425127
- [Background] Becher E, Roehrborn CG, Siami P, Gagnier RP, Wilson TH, Montorsi F. The effects of dutasteride, tamsulosin, and the combination on storage and voiding in men with benign prostatic hyperplasia and prostatic enlargement: 2-year results from the Combination of Avodart and Tamsulosin study. Prostate Cancer Prostatic Dis. 2009;12(4):369-74. doi: 10.1038/pcan.2009.37. Epub 2009 Sep 1. PMID 19901936
- [Background] Montorsi F, Roehrborn C, Garcia-Penit J, Borre M, Roeleveld TA, Alimi JC, Gagnier P, Wilson TH. The effects of dutasteride or tamsulosin alone and in combination on storage and voiding symptoms in men with lower urinary tract symptoms (LUTS) and benign prostatic hyperplasia (BPH): 4-year data from the Combination of Avodart and Tamsulosin (CombAT) study. BJU Int. 2011 May;107(9):1426-31. doi: 10.1111/j.1464-410X.2011.10129.x. Epub 2011 Feb 23. PMID 21348912
- [Background] Montorsi F, Henkel T, Geboers A, Mirone V, Arrosagaray P, Morrill B, Black L. Effect of dutasteride, tamsulosin and the combination on patient-reported quality of life and treatment satisfaction in men with moderate-to-severe benign prostatic hyperplasia: 4-year data from the CombAT study. Int J Clin Pract. 2010 Jul;64(8):1042-51. doi: 10.1111/j.1742-1241.2010.02428.x. Epub 2010 May 7. PMID 20487046
- [Background] Haillot O, Fraga A, Maciukiewicz P, Pushkar D, Tammela T, Hofner K, Chantada V, Gagnier P, Morrill B. The effects of combination therapy with dutasteride plus tamsulosin on clinical outcomes in men with symptomatic BPH: 4-year post hoc analysis of European men in the CombAT study. Prostate Cancer Prostatic Dis. 2011 Dec;14(4):302-6. doi: 10.1038/pcan.2011.13. Epub 2011 Apr 19. PMID 21502969
- [Background] Roehrborn CG, Siami P, Barkin J, Damiao R, Major-Walker K, Morrill B, Montorsi F; CombAT Study Group. The effects of dutasteride, tamsulosin and combination therapy on lower urinary tract symptoms in men with benign prostatic hyperplasia and prostatic enlargement: 2-year results from the CombAT study. J Urol. 2008 Feb;179(2):616-21; discussion 621. doi: 10.1016/j.juro.2007.09.084. Epub 2007 Dec 21. PMID 18082216
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: ARI40005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ARI40005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ARI40005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ARI40005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ARI40005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ARI40005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ARI40005 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In a 4-week, single-blind placebo run-in period, all participants (par.) took two capsules consisting of one dutasteride-matched placebo capsule and one tamsulosin-matched placebo capsule once daily for 4 weeks. A safety follow-up was performed for all participants 16 weeks after the last dose of study drug.
Groups:
- Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg: Dutasteride 0.5 milligrams (mg) plus tamsulosin 0.4 mg once daily for 208 weeks
- Dutasteride 0.5 mg: Dutasteride 0.5 mg plus tamsulosin placebo once daily for 208 weeks
- Tamsulosin 0.4 mg: Tamsulosin 0.4 mg plus dutasteride placebo once daily for 208 weeks
Period: Four-Year Double-Blind Treatment Period
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Started | 1610 | 1623 | 1611
Completed | 1113 | 1093 | 989
Not Completed | 497 | 530 | 622
Not completed — Adverse Event | 211 | 185 | 210
Not completed — Withdrawal by Subject | 114 | 160 | 148
Not completed — Lost to Follow-up | 53 | 48 | 58
Not completed — Protocol Violation | 29 | 29 | 34
Not completed — Lack of Efficacy | 53 | 71 | 104
Not completed — Participant Relocated | 7 | 2 | 8
Not completed — Site Closed/Sponsor Termination | 7 | 7 | 4
Not completed — Non-compliant/Medication Interruption | 6 | 4 | 7
Not completed — Prostate Surgery/TURP/Alt. Therapy | 3 | 7 | 19
Not completed — Participant Decision/Withdrawn | 2 | 0 | 4
Not completed — Acute Urinary Retention (AUR) | 2 | 3 | 6
Not completed — Prohibited Medication | 2 | 2 | 8
Not completed — Investigator Departure | 2 | 0 | 0
Not completed — Alcohol Dependent | 1 | 0 | 0
Not completed — Screen Failure | 1 | 0 | 0
Not completed — No Improvement | 1 | 0 | 0
Not completed — BPH/BPH symptoms worse/urinary incont. | 1 | 0 | 5
Not completed — Financial Problems | 1 | 0 | 0
Not completed — Loss of Libido | 1 | 0 | 0
Not completed — Angina Pectoris | 0 | 2 | 0
Not completed — Loss of Contact | 0 | 1 | 0
Not completed — Neoplasm of Bladder/Prostate | 0 | 1 | 1
Not completed — Cardiologist/Neurologist Decision | 0 | 2 | 0
Not completed — Renal Insufficiency | 0 | 1 | 0
Not completed — Back Pain | 0 | 1 | 0
Not completed — Scheduling Issues | 0 | 1 | 0
Not completed — Any Appreciable Improvement | 0 | 1 | 0
Not completed — Investigator Decision | 0 | 1 | 3
Not completed — Enrollment Error | 0 | 0 | 2
Not completed — Urinary Tract Infection (UTI) | 0 | 0 | 1
Not completed — Prostate Specific Antigen Rising | 0 | 1 | 0
Period: 16-Week Safety Follow-up Period
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Started | 1598 (Some par. didn't enter the Follow-up phase or dropped out before completing the treatment phase.) | 1615 (Some par. didn't enter the Follow-up phase or dropped out before completing the treatment phase.) | 1600 (Some par. didn't enter the Follow-up phase or dropped out before completing the treatment phase.)
Completed | 1224 | 1205 | 1143
Not Completed | 374 | 410 | 457
Not completed — Adverse Event | 34 | 39 | 44
Not completed — Withdrawal by Subject | 185 | 212 | 229
Not completed — Lost to Follow-up | 101 | 97 | 111
Not completed — Protocol Violation | 18 | 18 | 17
Not completed — Site Closed/Sponsor Termination | 8 | 5 | 4
Not completed — Non-compliant/Medication Interruption | 8 | 6 | 4
Not completed — Loss of Contact | 4 | 0 | 2
Not completed — Disease Progression/Treatment Failure | 3 | 1 | 1
Not completed — Participant relocated | 2 | 3 | 1
Not completed — Participant Decision/Withdrawn | 2 | 1 | 2
Not completed — Prohibited Medication | 2 | 3 | 5
Not completed — Alcohol Dependent | 1 | 0 | 1
Not completed — Prostate surgery/TURP/Alt. therapy | 1 | 5 | 13
Not completed — Loss of Libido | 1 | 0 | 0
Not completed — Enrollment Error | 1 | 0 | 2
Not completed — Neoplasm of Bladder/Prostate Cancer | 1 | 3 | 6
Not completed — Death | 1 | 0 | 1
Not completed — Gyneomastia | 1 | 0 | 0
Not completed — Acute Urinary Retention (AUR) | 0 | 5 | 4
Not completed — BPH/BPH symptoms worse/urinary incont. | 0 | 2 | 3
Not completed — Angina Pectoris | 0 | 1 | 0
Not completed — Back Pain | 0 | 1 | 0
Not completed — Scheduling Issues | 0 | 2 | 4
Not completed — Investigator/Sponsor Decision | 0 | 2 | 3
Not completed — Depression | 0 | 1 | 0
Not completed — Diabetes Uncontrolled | 0 | 1 | 0
Not completed — Jailed | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg | Total
Number analyzed (Participants) | 1610 | 1623 | 1611 | 4844
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (7.05) | 66.0 (6.99) | 66.2 (7.00) | 66.1 (7.01)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 1610 | 1623 | 1611 | 4844
Race/Ethnicity, Customized [Number; unit: participants]
  White | 1421 | 1433 | 1405 | 4259
  Black | 22 | 17 | 24 | 63
  Asian | 107 | 106 | 112 | 325
  American Hispanic | 44 | 48 | 55 | 147
  Unknown | 16 | 19 | 15 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Events of Acute Urinary Retention (AUR) or Benign Prostatic Hyperplasia (BPH)-Related Prostatic Surgery at the Indicated Time Periods.
Description: A participant was considered to have AUR when he was unable to urinate and required bladder catheterization. BPH is also known as an enlarged prostate. When symptoms of BPH become bothersome, surgery may be required. When events of AUR and BPH-related surgery were participant-reported or identified, they were recorded in the participants' clinic record.
Time Frame: Years 1, 2, 3, and 4
Population: Intent-to-Treat (ITT) Population: all participants randomized to the double-blind treatment period. As the study progressed, participants dropped out of the study.
Measure: Number; unit: events
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1610 | 1623 | 1611
events
  Year 1, n=1610, 1623, 1611 | 29 | 27 | 40
  Year 2, n=1457, 1484, 1464 | 14 | 22 | 62
  Year 3, n=1347, 1365, 1307 | 15 | 16 | 44
  Year 4, n=1274, 1277, 1176 | 9 | 19 | 45
Statistical Analysis 1: Comparison: Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.18, Log Rank — Log-rank test with stratification by cluster; Relative Risk Estimate = 0.80, 95% CI [0.58 to 1.11]
Statistical Analysis 2: Comparison: Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p < 0.001, Log Rank — Log-rank test with stratification by cluster; Relative Risk Estimate = 0.34, 95% CI [0.26 to 0.45]

2. Secondary Outcome: Number of Events of First BPH Clinical Progression at Years 1, 2, 3 and 4
Description: The time when the first symptom/event of BPH clinical progression has occurred (i.e. AUR, incontinence) was measured. Summaries are based on the first occuring event after treatment start. The time period is from treatment start to each participant's last treatment visit. The Year 4 events include all those that occur during the fourth year and beyond.
Time Frame: Years 1, 2, 3, and 4
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Number; unit: events
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1610 | 1623 | 1611
events
  Year 1, n=1610, 1623, 1611 | 126 | 184 | 171
  Year 2, n= 1264, 1240, 1262 | 31 | 54 | 78
  Year 3, n=1135, 1082, 1048 | 30 | 29 | 67
  Year 4, n= 1047, 959, 880 | 16 | 22 | 31

3. Primary Outcome: Number of Participants With AUR or BPH-related Surgery
Description: A participant was considered to have AUR when he was unable to urinate and required bladder catheterization. BPH is also known as an enlarged prostate. When symptoms of BPH become bothersome, surgery may be required. When events of AUR and BPH-related surgery were participant reported or identified, they were recorded in the participants' clinic record.
Time Frame: Baseline (Day 1) through Year 4
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1610 | 1623 | 1611
participants
  AUR | 35 | 44 | 109
  BPH-related surgery | 32 | 40 | 82
Statistical Analysis 1: Comparison: Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.18, Log Rank — Log rank test with stratification by cluster
Statistical Analysis 2: Comparison: Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p < 0.001, Log Rank — Log rank test with stratification by cluster

4. Secondary Outcome: The Number of Participants With Each of the Five Components of BPH Clinical Progression
Description: The five components measured were symptom deterioration, BPH-related AUR, BPH-related incontinence, recurrent BPH-related Urinary Tract Infection (UTI), and BPH-related renal insufficiency.
Time Frame: Baseline (Day 1) to Year 4
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1610 | 1623 | 1611
participants
  Symptom deterioration | 132 | 203 | 221
  BPH-related AUR | 22 | 31 | 64
  BPH-related incontinence | 46 | 49 | 56
  Recurrent BPH-related UTI | 2 | 5 | 3
  BPH-related renal insufficiency | 1 | 2 | 5

5. Secondary Outcome: Number of Events of Symptom Deterioration at the Indicated Time Periods
Description: The number of participants (par.) with symptom deterioration of International Prostate Symptom Score (IPSS) ≥4 points on two consecutive visits post-baseline are presented. Data are based on the first occurrence of an event after treatment start. The year-4 events include all that occured during the 4th year and beyond. The IPSS is a 7-item questionnaire measuring the level of urinary symptoms reported as the total score. Each question has a 6-point response scale (0=none/not at all to 5=almost always), with a total score ranging from 0-35: mild (0-7), moderate (8-19), or severe (20-35).
Time Frame: Years 1, 2, 3, and 4 (from treatment start until each participant's last treatment-phase visit)
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1610 | 1623 | 1611
events
  Year 1, n=1610, 1623, 1611 | 91 | 138 | 119
  Year 2, n=1286, 1278, 1296 | 23 | 38 | 49
  Year 3, n=1158, 1132, 1088 | 14 | 23 | 42
  Year 4, n=1083, 1001, 926 | 11 | 13 | 19
Statistical Analysis 1: Comparison: Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg vs Dutasteride 0.5 mg; Test type: Superiority or Other; p < 0.001, Log Rank; Log-rank test with stratification by cluster; Relative Risk Estimate = 0.65, 95% CI [0.52 to 0.80]
Statistical Analysis 2: Comparison: Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p < 0.001, Log Rank; Relative Risk Estimate = 0.59, 95% CI [0.48 to 0.72]

6. Secondary Outcome: Number of Participants With an Event of Post-baseline BPH-related Macroscopic Hematuria
Description: A participant was considered to have macroscopic hematuria when there was presence of blood in the urine. The event of macroscopic hematuria was either participant-reported or identified by the investigator during a clinic visit. Overall Crude Rate is the number of participants from the total number analyzed that experience experienced an incident of post-baseline BPH or Non-BPH related macroscopic hematuria. Participants may appear in both categories.
Time Frame: Baseline (Day 1) through Year 4
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1610 | 1623 | 1611
participants
  Overall crude rate | 53 | 70 | 81
  Non-BPH-related Crude Rate | 15 | 28 | 25
  BPH-Related Crude Rate | 40 | 45 | 56
Statistical Analysis 1: Comparison: Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.65, Log Rank; Mantel-Haenszel test with stratification by cluster
Statistical Analysis 2: Comparison: Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.10, Log Rank; Mantel-Hanenszel test with stratification by cluster

7. Secondary Outcome: Number of Participants With an Event of Post-baseline BPH-related Hematospermia
Description: A participant was considered to have hematospermia when there was presence of blood in the semen. Hematospermia can occur from prostatitis (prostate infection), from cancer, or after a prostate biopsy. The event of hematospermia was either participant-reported or identified by the investigator during a clinic visit. Overall Crude Rate is the number of participants from the total number analyzed that experience experienced an incident of post-baseline BPH or Non-BPH related hematospermia. Participants may appear in both categories.
Time Frame: Baseline (Day 1) through Year 4
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1610 | 1623 | 1611
participants
  Overall Crude Rate | 18 | 19 | 20
  Non-BPH-related Crude Rate | 2 | 3 | 9
  BPH-related Crude Rate | 17 | 17 | 11
Statistical Analysis 1: Comparison: Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg vs Dutasteride 0.5 mg; Test type: Superiority or Other; p = 0.95, Log Rank; Mantel-Haenszel test with stratification by cluster
Statistical Analysis 2: Comparison: Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg vs Tamsulosin 0.4 mg; Test type: Superiority or Other; p = 0.24, Log Rank; Mantel-Haenszel test with stratification by cluster

8. Secondary Outcome: Adjusted Mean Change From Baseline in International Prostate Symptom Score (IPSS) at Months 12, 24, 36, and 48
Description: The IPSS is a 7-item questionnaire that measures urinary symptoms. It measures the level of urinary symptoms (including incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia) reported as the total IPSS score. Each of the 7 questions has a 6-point response scale (0=none/not at all to 5=almost always) with a total score that can range from 0-35: mild (0-7), moderate (8-19), or severe (20-35). Estimates are based on adjusted (least squares) means from the general linear model: change from baseline IPSS = Treatment + Cluster + Baseline IPSS.
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1575 | 1592 | 1582
points on a scale
  Month 12 | -5.6 (0.15) | -4.2 (0.15) | -4.5 (0.15)
  Month 24 | -6.2 (0.15) | -4.9 (0.15) | -4.3 (0.15)
  Month 36 | -6.3 (0.16) | -5.2 (0.16) | -4.0 (0.16)
  Month 48 | -6.3 (0.16) | -5.3 (0.16) | -3.8 (0.16)

9. Secondary Outcome: Adjusted Mean Change From Baseline in Urinary Flow Rate (Qmax) at Months 12, 24, 36, and 48
Description: Peak maximum urinary flow (Qmax) of urinary flow using a Medtronic (formerly Dantec) Uroflow Meter (Urodyn 1000 or Duet models) with a Thompson filter was measured. Estimates are based on adjusted (least squares) means from the general linear model: Change from baseline Qmax = treatment + cluster + baseline Qmax.
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: ITT Population. As the study progressed, participants dropped out of the study. Also, assessments with voided volumes <125 ml were not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: milliliters (mL)/second (sec)
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1495 | 1505 | 1523
milliliters (mL)/second (sec)
  Month 12, n=1477, 1482, 1510 | 2.0 (0.12) | 1.5 (0.12) | 0.9 (0.12)
  Month 24, n= 1492, 1501, 1519 | 2.4 (0.12) | 1.9 (0.12) | 0.9 (0.12)
  Month 36, n= 1495, 1504, 1521 | 2.6 (0.12) | 1.9 (0.12) | 0.6 (0.12)
  Month 48, n= 1495, 1505, 1523 | 2.4 (0.13) | 2.0 (0.13) | 0.7 (0.13)

10. Secondary Outcome: Adjusted Mean Percent Change From Baseline in Prostate Volume at Months 12, 24, 36, and 48
Description: Prostate volume measurements were conducted annually using Transurethral ultrasound (TRUS). The anteroposterior, cephalocaudal, and transverse diameters of the prostate obtained by TRUS calculate the total prostate volume centimeters (cc). Percent change from baseline = [(post-baseline - baseline)/baseline value] x 100. Estimates were based on the adjusted (least squares) means from the general linear model: log(post-baseline/baseline value) + treatment + cluster + log(baseline value) and are reported as percent change from baseline.
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: ITT Population. As the study progressed, participants dropped out of the study. Also, prostate measurements were either not performed or missing for some participants at various timepoints.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1430 | 1455 | 1468
percent change
  Month 12, n=1411, 1442, 1451 | -24.1 (0.60) | -25.2 (0.59) | -1.5 (0.77)
  Month 24, n= 1427, 1451, 1465 | -26.9 (0.62) | -28.0 (0.61) | 0.0 (0.84)
  Month 36, n= 1430, 1455, 1468 | -27.6 (0.68) | -28.8 (0.66) | 1.6 (0.94)
  Month 48, n= 1430, 1455, 1468 | -27.3 (0.66) | -28.0 (0.65) | 4.6 (0.94)

11. Secondary Outcome: Adjusted Mean Change From Baseline in Transition Zone (Portion of the Prostate That Surrounds the Proximal Urethra) Volume at Months 12, 24, 36, and 48
Description: Prostate volume (PV) measurements were conducted annually using Transurethral ultrasound (TRUS). The anteroposterior, cephalocaudal, and transverse diameters of the prostate obtained by TRUS calculate the total PV in centimeters (cc). Results are for the transition zone measurements of the prostate in a small subset of participants. Percent change from baseline (BL) = [(post-BL - BL)/BL value] x 100. Estimates are based on the adjusted (least squares) means for the general linear model: log(post-BL/BL value) = treatment + cluster + log(BL value) and are reported as percent change from BL.
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: ITT Population. As the study progressed, participants dropped out of the study. Transition zone measurements were only done on a subset of participants at sites with experience in measuring the transition zone of the prostate. Also, transition zone measurements were either not performed or missing for some participants at various timepoints.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 155 | 164 | 163
percent change
  Month 12, n= 150, 159, 160 | -17.2 (3.29) | -15.6 (3.39) | 5.6 (4.09)
  Month 24, n= 153, 164, 160 | -23.4 (5.63) | -22.8 (5.86) | 8.7 (8.22)
  Month 36, n= 155, 164, 162 | -20.9 (3.97) | -26.7 (3.90) | 14.7 (5.89)
  Month 48, n= 155, 164, 163 | -17.9 (4.45) | -26.5 (4.21) | 18.2 (6.54)

12. Secondary Outcome: Number of Unscheduled Visits to GP/Urologist Regarding AUR Symptoms Since the Last Study Visit
Description: At each scheduled 13-week clinic visit post-randomization, the investigator was to record details of any health care utilization associated with an episode of AUR. Responses to the following question were recorded: "Has the participant needed to make any unscheduled visits to his general practitioner (GP)/Urologist regarding AUR symptoms since the last study visit?" If the answer to the question was "yes," the number of visits was recorded.
Time Frame: Every 3 months from Month 3 to Month 48
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Number; unit: visits
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1550 | 1581 | 1565
visits
  Month 3, n=1550, 1581, 1565 | 8 | 6 | 7
  Month 6, n=1479, 1517, 1514 | 2 | 4 | 3
  Month 9, n=1439, 1465, 1477 | 4 | 3 | 8
  Month 12, n=1400, 1431, 1434 | 3 | 3 | 9
  Month 15, n=1343, 1386, 1380 | 3 | 6 | 6
  Month 18, n=1318, 1350, 1328 | 3 | 4 | 10
  Month 21, n=1281, 1326, 1287 | 3 | 3 | 9
  Month 24, n=1263, 1293, 1244 | 2 | 2 | 7
  Month 27, n=1233, 1262, 1206 | 1 | 6 | 7
  Month 30, n=1222, 1221, 1166 | 3 | 2 | 8
  Month 33, n=1202, 1199, 1128 | 3 | 4 | 5
  Month 36, n=1187, 1174, 1095 | 2 | 1 | 5
  Month 39, n=1160, 1144, 1055 | 2 | 2 | 5
  Month 42, n=1149, 1126, 1035 | 3 | 2 | 8
  Month 45, n=1129, 1110, 1009 | 1 | 2 | 4
  Month 48, n=1113, 1093, 990 | 1 | 2 | 2

13. Secondary Outcome: Number of "Yes" Responses to the Question: "Would the Participant Have Paid a Visit to His GP/Urologist Regarding AUR Symptoms if the Study Visit Had Not Been Planned"?.
Description: At each scheduled 13-week clinic visit post-randomization, the investigator was to record details of any health care utilization associated with an episode of AUR. Responses to the following question were recorded: "Would the participant have paid a visit to his GP/Urologist regarding AUR symptoms if this study visit had not been planned?". If the answer to the question was "yes," the number of Yes responses was recorded.
Time Frame: Every 3 months from Month 3 to Month 48
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Number; unit: yes responses
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1550 | 1581 | 1564
yes responses
  Month 3, n=1550, 1581, 1564 | 31 | 32 | 29
  Month 6, n=1479, 1516, 1513 | 21 | 26 | 26
  Month 9, n=1439, 1465, 1477 | 18 | 14 | 18
  Month 12, n=1400, 1431, 1434 | 8 | 13 | 9
  Month 15, n=1343, 1386, 1380 | 9 | 15 | 12
  Month 18, n=1318, 1350, 1328 | 17 | 13 | 19
  Month 21, n=1281, 1326, 1287 | 10 | 15 | 17
  Month 24, n=1263, 1293, 1244 | 5 | 9 | 8
  Month 27, n=1233, 1262, 1206 | 9 | 11 | 8
  Month 30, n=1222, 1221, 1166 | 7 | 9 | 9
  Month 33, n=1202, 1199, 1128 | 9 | 10 | 11
  Month 36, n=1187, 1174, 1095 | 5 | 4 | 5
  Month 39, n=1160, 1144, 1055 | 7 | 9 | 6
  Month 42, n=1149, 1126, 1035 | 6 | 8 | 8
  Month 45, n=1129, 1110, 1009 | 7 | 8 | 5
  Month 48, n=1113, 1093, 990 | 2 | 9 | 5

14. Secondary Outcome: Number of Visits to GP/Urologist Regarding BPH-related Surgery Since the Last Study Visit
Description: At each scheduled 13-week clinic visit post-randomization, the investigator was to record details of any health care utilization associated with BPH-related surgery. Responses to the following question were recorded: "Has the participant needed to visit his general practitioner (GP)/Urologist regarding BPH-related surgery since the last study visit?". If the answer to the question was "yes," the number of visits was recorded.
Time Frame: Every 3 months from Month 3 to Month 48
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Number; unit: visits
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1550 | 1581 | 1564
visits
  Month 3, n=1550, 1581, 1564 | 0 | 3 | 3
  Month 6, n=1479, 1517, 1514 | 2 | 1 | 2
  Month 9, n=1439, 1465, 1477 | 2 | 2 | 3
  Month 12, n=1400, 1431, 1434 | 1 | 2 | 7
  Month 15, n=1343, 1386, 1380 | 2 | 5 | 7
  Month 18, n=1318, 1350, 1328 | 4 | 0 | 4
  Month 21, n=1281, 1326, 1287 | 1 | 0 | 3
  Month 24, n=1263, 1293, 1244 | 2 | 0 | 3
  Month 27, n=1233, 1262, 1206 | 3 | 3 | 4
  Month 30, n=1222, 1221, 1165 | 0 | 1 | 1
  Month 33, n=1202, 1199, 1128 | 0 | 1 | 5
  Month 36, n=1187, 1174, 1095 | 2 | 2 | 1
  Month 39, n=1160, 1144, 1055 | 1 | 3 | 2
  Month 42, n=1149, 1126, 1035 | 1 | 2 | 5
  Month 45, n=1129, 1110, 1009 | 0 | 3 | 2
  Month 48, n=1113, 1093, 990 | 0 | 2 | 1

15. Secondary Outcome: Number of "Yes" Responses to the Question: "Would the Participant Have Paid a Visit to His GP/Urologist Regarding BPH-related Surgery Since the Last Study Visit?"
Description: At each scheduled 13-week clinic visit post-randomization, the investigator was to record details of any health care utilization associated with BPH-related surgery. Responses to the following question were recorded: "Would the participant have paid a visit to his general practitioner (GP)/Urologist regarding BPH-related surgery since the last study visit?". If the answer to the question was "yes," the number of Yes responses was recorded.
Time Frame: Every 3 months from Month 3 to Month 48
Population: ITT Population. As study progressed, participants dropped out of study.
Measure: Number; unit: yes responses
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1550 | 1581 | 1564
yes responses
  Month 3, n=1550, 1581, 1564 | 16 | 34 | 28
  Month 6, n=1479, 1516, 1513 | 20 | 23 | 16
  Month 9, n=1438, 1465, 1477 | 12 | 10 | 17
  Month 12, n=1400, 1431, 1434 | 5 | 10 | 6
  Month 15, n=1343, 1386, 1380 | 9 | 9 | 9
  Month 18, n=1318, 1350, 1328 | 13 | 12 | 10
  Month 21, n=1281, 1326, 1287 | 10 | 9 | 8
  Month 24, n=1263, 1293, 1244 | 4 | 7 | 3
  Month 27, n=1233, 1262, 1206 | 9 | 9 | 5
  Month 30, n=1222, 1221, 1166 | 7 | 9 | 4
  Month 33, n=1202, 1199, 1128 | 5 | 7 | 8
  Month 36, n=1187, 1174, 1095 | 3 | 5 | 2
  Month 39, n=1160, 1144, 1055 | 7 | 8 | 5
  Month 42, n=1149, 1126, 1034 | 9 | 8 | 2
  Month 45, n=1129, 1110, 1009 | 6 | 8 | 5
  Month 48, n=1113, 1093, 990 | 1 | 3 | 1

16. Secondary Outcome: Number of Unplanned Visits to GP/Urologist That Would Have Taken Place if a Scheduled Study Visit Had Not Been Planned (Including Visits Resulting From UTI, UI, Macroscopic Haematuria, Etc.)
Description: At each scheduled 13-week clinic visit post-randomization, the investigator was to record details of any health care utilization associated with unplanned visits to GP/Urologist. Responses to the following question were recorded: "Has the participant had any unplanned GP/Urologist (outpatient) visits that would have taken place if a scheduled study visit had not been planned (this can include visits resulting from UTI, UI macroscopic haematuria, etc?". If the answer to the question was "yes," the number of visits was recorded.
Time Frame: Every 3 months from Month 3 to Month 48
Population: ITT Population. As study progressed, participants dropped out of the study.
Measure: Number; unit: visits
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1550 | 1581 | 1564
visits
  Month 3, n=1550, 1581, 1564 | 23 | 25 | 26
  Month 6, n=1479, 1517, 1514 | 23 | 34 | 22
  Month 9, n=1439, 1465, 1477 | 16 | 35 | 22
  Month 12, n=1400, 1431, 1434 | 30 | 29 | 34
  Month 15, n=1343, 1386, 1380 | 24 | 22 | 27
  Month 18, n=1318, 1350, 1328 | 21 | 25 | 26
  Month 21, n=1281, 1326, 1287 | 18 | 21 | 14
  Month 24, n=1263, 1293, 1244 | 10 | 19 | 21
  Month 27, n=1233, 1262, 1206 | 15 | 11 | 14
  Month 30, n=1222, 1221, 1166 | 7 | 8 | 10
  Month 33, n=1202, 1199, 1128 | 4 | 5 | 10
  Month 36, n=1187, 1174, 1095 | 5 | 4 | 7
  Month 39, n=1160, 1144, 1055 | 6 | 13 | 19
  Month 42, n=1149, 1126, 1035 | 4 | 8 | 12
  Month 45, n=1129, 1110, 1009 | 3 | 5 | 6
  Month 48, n=1113, 1093, 990 | 1 | 6 | 5

17. Secondary Outcome: Number of Unscheduled Visits to GP/Urologist (Outpatient) Planned, Not Relating to the Study (Including Visits Resulting From UTI, UI, Macroscopic Haematuria, Etc.)
Description: At each scheduled 13-week clinic visit post-randomization, the investigator was to record details of any health care utilization associated with unplanned visits to GP/Urologist. Responses to the following question were recorded: "Does the participant have any unscheduled GP/Urologist (outpatients) visits planned, not relating to the study (this can include visits resulting from UTI, UI, macroscopic haematuria, etc.?". If the answer to the question was "yes," the number of visits was recorded.
Time Frame: Every 3 months from Month 3 to Month 48
Population: ITT Population. As study progressed, participants dropped out the study.
Measure: Number; unit: visits
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1550 | 1581 | 1564
visits
  Month 3, n=1550, 1581, 1564 | 27 | 27 | 30
  Month 6, n=1479, 1516, 1514 | 23 | 29 | 33
  Month 9, n=1439, 1465, 1477 | 12 | 27 | 26
  Month 12, n=1400, 1431, 1434 | 30 | 28 | 29
  Month 15, n=1343, 1386, 1381 | 19 | 28 | 32
  Month 18, n=1318, 1350, 1328 | 23 | 21 | 34
  Month 21, n=1281, 1326, 1287 | 20 | 27 | 26
  Month 24, n=1263, 1293, 1244 | 29 | 23 | 26
  Month 27, n=1233, 1262, 1206 | 13 | 12 | 16
  Month 30, n=1222, 1221, 1166 | 10 | 16 | 10
  Month 33, n=1202, 1199, 1128 | 6 | 13 | 20
  Month 36, n=1187, 1174, 1095 | 8 | 12 | 18
  Month 39, n=1160, 1144, 1055 | 12 | 10 | 18
  Month 42, n=1149, 1126, 1035 | 15 | 9 | 15
  Month 45, n=1129, 1110, 1009 | 5 | 7 | 8
  Month 48, n=1113, 1093, 990 | 7 | 4 | 8

18. Secondary Outcome: Adjusted Mean Change From Baseline in BPH Impact Index (BII) at Months 12, 24, 36, and 48
Description: The BII is a 4-item questionnaire, score range of 0 (best) to 12 (worst) for questions 1-3, and 0 (best) to 13 (worst) for question 4, that assesses the overall impact of BPH on a participant's general sense of well being and measures aspects of physical discomfort, worry, and bother, all of which can be affected by BPH and its symptoms. BII score = sum of questions 1-4. Change from baseline = Post-Baseline Value. Estimates are based on the adjusted (least squares) means from the general linear model: change from baseline BII = treatment + cluster + baseline BII.
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1574 | 1593 | 1582
points on a scale
  Month 12 | -1.9 (0.06) | -1.5 (0.06) | -1.6 (0.06)
  Month 24 | -2.1 (0.07) | -1.7 (0.07) | -1.5 (0.07)
  Month 36 | -2.2 (0.07) | -1.8 (0.07) | -1.3 (0.07)
  Month 48 | -2.2 (0.07) | -1.8 (0.07) | -1.2 (0.07)

19. Secondary Outcome: Adjusted Mean Change From Baseline in BPH-Related Health Status (BHS) at Months 12, 24, 36, and 48
Description: The effect of study treatment on BHS was assessed by using three self-administered questionnaires: the International Prostate Symptom Score (IPSS), the BPH Impact Index (BII), and Patient Perception of Study Medication (PPSM). The BHS score was collected on the IPPS questionnaire and ranged from 0 (best) to 6 (worst). Percent change from baseline = [(post-baseline - baseline)/baseline value] x 100. Estimates were based on the adjusted (least squares) means from the general linear model: change from baseline BPH-related health status = treatment + cluster + baseline BPH-Related health status.
Time Frame: Baseline and Months 12, 24, 36, 48
Population: ITT Population. As the study progressed, participants dropped out of the study.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1575 | 1592 | 1583
points on a scale
  Month 12 | -1.2 (0.03) | -1.0 (0.03) | -1.0 (0.03)
  Month 24 | -1.4 (0.03) | -1.1 (0.03) | -1.1 (0.03)
  Month 36 | -1.5 (0.03) | -1.2 (0.03) | -1.1 (0.03)
  Month 48 | -1.5 (0.03) | -1.3 (0.03) | -1.1 (0.03)

20. Secondary Outcome: Patient Perception of Study Medication (PPSM): Number of Participants With the Indicated Responses to Question 1 (LOCF)
Description: This 12-item questionnaire (PPSM) was developed by GlaxoSmithKline for use in this study and was designed to quantify the participant's perceptions and satisfaction with the effect of study treatment on control of their urinary symptoms at baseline and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and 48. Participants were asked to respond to the question of "Since you began taking the study medication, how has control of your urinary problems changed?".
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: ITT Population. As the study progressed, participants dropped out of the study. Only participants responding to the question were analyzed.
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1685 | 1600 | 1586
participants
  Baseline (BL), Any Improvement, n=1585, 1600, 1586 | 696 | 656 | 706
  BL, No Change/Any Worsening, n=1585, 1600, 1586 | 889 | 944 | 880
  Month (M) 12, Any Improvement, n=1576, 1593, 1581 | 1281 | 1171 | 1218
  M12, No Change/Any Worsening, n=1576, 1593, 1581 | 295 | 422 | 363
  M24, Any Improvement, n=1576, 1593, 1581 | 1273 | 1200 | 1195
  M24, No Change/Any Worsening, n=1576, 1593, 1581 | 303 | 393 | 386
  M36, Any Improvement, n=1576, 1593, 1581 | 1268 | 1203 | 1152
  M36, No Change/Any Worsening, n=1576, 1593, 1581 | 308 | 390 | 429
  M48, Any Improvement, n=1576, 1593, 1581 | 1278 | 1212 | 1138
  M48, No Change/Any Worsening, n=1576, 1593, 1581 | 298 | 381 | 443

21. Secondary Outcome: Patient Perception of Study Medication (PPSM): Number of Participants With the Indicated Responses to Question 2 (LOCF)
Description: This 12-item questionnaire (PPSM) was developed by GlaxoSmithKline for use in this study and was designed to quantify the participant's perceptions and satisfaction with the effect of study treatment on control of their urinary symptoms at baseline and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and 48. Participants were asked to respond to the question of "How satisfied are you with the effect of the study medication on control of your urinary problems?" Satisfact., satisfaction.
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1587 | 1600 | 1583
participants
  Baseline (BL), Any Satisfact., n=1587, 1600, 1583 | 707 | 652 | 686
  BL, Neutral/Any Dissatisfact., n=1587, 1600, 1583 | 880 | 948 | 897
  Month (M) 12, Any Satisfact., n=1576, 1593, 1581 | 1224 | 1127 | 1178
  M12, Neutral/Any Dissatisfact., n=1576, 1593, 1581 | 352 | 466 | 403
  M24, Any Satisfact., n=1576, 1593, 1581 | 1261 | 1166 | 1150
  M24, Neutral/Any Dissatisfact., n=1576, 1593, 1581 | 315 | 427 | 431
  M36, Any Satisfact., n=1576, 1593, 1581 | 1260 | 1167 | 1120
  M36, Neutral/Any Dissatisfact., n=1576, 1593, 1581 | 316 | 426 | 461
  M48, Any Satisfact., n=1576, 1593, 1581 | 1267 | 1172 | 1088
  M48, Neutral/Any Dissatisfact., n=1576, 1593, 1581 | 309 | 421 | 493

22. Secondary Outcome: Patient Perception of Study Medication (PPSM): Number of Participants With the Indicated Responses to Question 3 (LOCF)
Description: This 12-item questionnaire (PPSM) was developed by GlaxoSmithKline for use in this study and was designed to quantify the participant's perceptions and satisfaction with the effect of study treatment on control of their urinary symptoms at baseline and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and 48. Participants were asked to respond to the question of "Since you began taking the study medication, how has the strength of your urinary stream changed?".
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1585 | 1601 | 1585
participants
  Baseline (BL), Any Improvement, n=1585, 1601, 1585 | 629 | 602 | 615
  BL, No Change/Any Worsening, n=1585, 1601, 1585 | 956 | 999 | 970
  Month (M) 12, Any Improvement, n=1576, 1593, 158 | 1181 | 1044 | 1105
  M12, No Change/Any Worsening, n=1576, 1593, 1581 | 395 | 549 | 476
  M24, Any Improvement, n=1576, 1593, 1581 | 1215 | 1070 | 1057
  M24, No Change/Any Worsening, n=1576, 1593, 1581 | 361 | 523 | 524
  M36, Any Improvement, n=1576, 1593, 1581 | 1206 | 1071 | 1023
  M36, No Change/Any Worsening, n=1576, 1593, 1581 | 370 | 522 | 558
  M48, Any Improvement, n=1576, 1593, 1581 | 1202 | 1086 | 1008
  M48, No Change/Any Worsening, n=1576, 1593, 1581 | 374 | 507 | 573

23. Secondary Outcome: Patient Perception of Study Medication (PPSM): Number of Participants With the Indicated Responses to Question 4 (LOCF)
Description: This 12-item questionnaire (PPSM) was developed by GlaxoSmithKline for use in this study and was designed to quantify the participant's perceptions and satisfaction with the effect of study treatment on control of their urinary symptoms at baseline and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and 48. Participants were asked to respond to the question of "How satisfied are you with the effect of the study medication on the strength of your urinary stream?". Satisfact., satisfaction.
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1583 | 1601 | 1582
participants
  Baseline (BL), Any Satisfact., n=1583,1601,1582 | 632 | 586 | 613
  BL, Neutral/Any Dissatisfact., n=1583,1601,1582 | 951 | 1015 | 969
  Month (M) 12, Any Satisfact., n=1576, 1593, 1581 | 1154 | 1037 | 1097
  M12, Neutral/Any Dissatisfact., n=1576, 1593, 1581 | 422 | 556 | 484
  M24, Any Satisfact., n=1576, 1593, 1581 | 1203 | 1072 | 1051
  M24, Neutral/Any Dissatisfact., n=1576, 1593, 1581 | 373 | 521 | 530
  M36, Any Satisfact., n=1576, 1593, 1581 | 1201 | 1075 | 1039
  M36, Neutral/Any Dissatisfact., n=1576, 1593, 1581 | 375 | 518 | 542
  M48, Any Satisfact., n=1576, 1593, 1581 | 1208 | 1089 | 1022
  M48, Neutral/Any Dissatisfact., n=1576, 1593, 1581 | 368 | 504 | 559

24. Secondary Outcome: Patient Perception of Study Medication (PPSM): Number of Participants With the Indicated Responses to Question 5 (LOCF)
Description: This 12-item questionnaire (PPSM) was developed by GlaxoSmithKline for use in this study and was designed to quantify the participant's perceptions and satisfaction with the effect of study treatment on control of their urinary symptoms at baseline and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and 48. Participants were asked to respond to the question of "Since you began taking the study medication, how has your pain prior to urinating changed?".
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 869 | 901 | 849
participants
  Baseline (BL), Any Improvement, n=869, 901, 849 | 337 | 331 | 332
  BL, No Change/Any Worsening, n=869, 901, 849 | 532 | 570 | 517
  Month (M) 12, Any Improvement, n=769, 817, 771 | 556 | 526 | 527
  M12, No Change/Any Worsening, n=769, 817, 771 | 213 | 291 | 244
  M24, Any Improvement, n=720, 780, 771 | 537 | 526 | 535
  M24, No Change/Any Worsening, n=720, 780, 771 | 183 | 254 | 236
  M36, Any Improvement, n=714, 753, 748 | 540 | 514 | 496
  M36, No Change/Any Worsening, n=714, 753, 748 | 174 | 239 | 252
  M48, Any Improvement, n=709, 756, 751 | 531 | 510 | 489
  M48, No Change/Any Worsening, n=709, 756, 751 | 178 | 246 | 262

25. Secondary Outcome: Patient Perception of Study Medication (PPSM): Number of Participants With the Indicated Responses to Question 6 (LOCF)
Description: This 12-item questionnaire (PPSM) was developed by GlaxoSmithKline for use in this study and was designed to quantify the participant's perceptions and satisfaction with the effect of study treatment on control of their urinary symptoms at baseline and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and 48. Participants were asked to respond to the question of "How satisfied are you with the effect the study medication has on your pain prior to urinating?". Satisfact., satisfaction.
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1135 | 1223 | 1161
participants
  Baseline (BL), Any Satisfact., n=908, 932, 889 | 375 | 351 | 351
  BL, Neutral/Any Dissatisfact., n=908, 932, 889 | 533 | 581 | 538
  Month (M) 12, Any Satisfact., n=1022, 1088, 1019 | 712 | 672 | 681
  M12, Neutral/Any Dissatisfact., n=1022, 1088, 1019 | 310 | 416 | 338
  M24, Any Satisfact., n=1077, 1151, 1085 | 764 | 740 | 708
  M24, Neutral/Any Dissatisfact., n=1077, 1151, 1085 | 313 | 411 | 377
  M36, Any Satisfact., n=1115, 1200, 1135 | 799 | 785 | 736
  M36, Neutral/Any Dissatisfact., n=1115, 1200, 1135 | 316 | 415 | 399
  M48, Any Satisfact., n=1135, 1223, 1161 | 810 | 792 | 739
  M48, Neutral/Any Dissatisfact., n=1135, 1223, 1161 | 325 | 431 | 422

26. Secondary Outcome: Patient Perception of Study Medication (PPSM): Number of Participants With the Indicated Responses to Question 7 (LOCF)
Description: This 12-item questionnaire (PPSM) was developed by GlaxoSmithKline for use in this study and was designed to quantify the participant's perceptions and satisfaction with the effect of study treatment on control of their urinary symptoms at baseline and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and 48. Participants were asked to respond to the question of "Since you began taking the study medication, how has your pain during urination changed?".
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 852 | 889 | 822
participants
  Baseline (BL), Any Improvement, n=852, 889, 822 | 321 | 314 | 319
  BL, No Change/Any Worsening, n=852, 889, 822 | 531 | 575 | 503
  Month (M) 12, Any Improvement, n=760, 781, 755 | 550 | 500 | 529
  M12, No Change/Any Worsening, n=760, 781, 755 | 210 | 281 | 226
  M24, Any Improvement, n=706, 760, 747 | 532 | 508 | 519
  M24, No Change/Any Worsening, n=706, 760, 747 | 174 | 252 | 228
  M36, Any Improvement, n=704, 741, 733 | 529 | 504 | 491
  M36, No Change/Any Worsening, n=704, 741, 733 | 175 | 237 | 242
  M48, No Change/Any Worsening, n=702, 739, 740 | 175 | 252 | 257
  M48, Any Improvement, n=702, 739, 740 | 527 | 487 | 483

27. Secondary Outcome: Patient Perception of Study Medication (PPSM): Number of Participants With the Indicated Responses to Question 8 (LOCF)
Description: This 12-item questionnaire (PPSM) was developed by GlaxoSmithKline for use in this study and was designed to quantify the participant's perceptions and satisfaction with the effect of study treatment on control of their urinary symptoms at baseline and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and 48. Participants were asked to respond to the question of "How satisfied are you with the effect the study medication has on your pain during urination?". Satisfact., satisfaction.
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1146 | 1224 | 1160
participants
  Baseline (BL), Any Satisfact., n=890, 925, 851 | 354 | 348 | 333
  BL, Neutral/Any Dissatisfact., n=890, 925, 851 | 536 | 577 | 518
  Month (M) 12, Any Satisfact., n=1022, 1088, 1011 | 712 | 655 | 678
  M12, Neutral/Any Dissatisfact., n=1022, 1088, 1011 | 310 | 433 | 333
  M24, Any Satisfact., n=1077, 1155, 1079 | 763 | 730 | 708
  M24, Neutral/Any Dissatisfact., n=1077, 1155, 1079 | 314 | 425 | 371
  M36, Any Satisfact., n=1121, 1206, 1131 | 807 | 784 | 724
  M36, Neutral/Any Dissatisfact., n=1121, 1206, 1131 | 314 | 422 | 407
  M48, Any Satsifact., n=1146,1224,1160 | 827 | 785 | 729
  M48, Neutral/Any Dissatisfact., n=1146, 1224, 1160 | 319 | 439 | 431

28. Secondary Outcome: Patient Perception of Study Medication (PPSM): Number of Participants With the Indicated Responses to Question 9 (LOCF)
Description: This 12-item questionnaire (PPSM) was developed by GlaxoSmithKline for use in this study and was designed to quantify the participant's perceptions and satisfaction with the effect of study treatment on control of their urinary symptoms at baseline and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and 48. Participants were asked to respond to the question of "Since you began taking the study medication, how has the way your urinary problems interfere with your ability to go about your usual activities changed?".
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1575 | 1593 | 1580
participants
  Baseline (BL), Any Improvement, n=1574, 1599, 1575 | 509 | 481 | 494
  BL, No Change/Any Worsening, n=1574, 1599, 1575 | 1065 | 1118 | 1081
  Month (M) 12, Any Improvement, n=1575, 1593, 1580 | 1124 | 1027 | 1084
  M12, No Change/Any Worsening, n=1575, 1593, 1580 | 451 | 566 | 496
  M24, Any Improvement, n=1575, 1593, 1580 | 1146 | 1053 | 1049
  M24, No Change/Any Worsening, n=1575, 1593, 1580 | 429 | 540 | 531
  M36, Any Improvement, n=1575, 1593, 1580 | 1575 | 1593 | 1580
  M36, No Change/Any Worsening, n=1575, 1593, 1580 | 412 | 529 | 553
  M48, Any Improvement, n=1575, 1593, 1580 | 1148 | 1063 | 1008
  M48, No Change/Any Worsening, n=1575, 1593, 1580 | 427 | 530 | 572

29. Secondary Outcome: Patient Perception of Study Medication (PPSM): Number of Participants With the Indicated Responses to Question 10 (LOCF)
Description: This 12-item questionnaire (PPSM) was developed by GlaxoSmithKline for use in this study and was designed to quantify the participant's perceptions and satisfaction with the effect of study treatment on control of their urinary symptoms at baseline and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and 48. Participants were asked to respond to the question of "How satisfied are you with the effect the study medication has on your ability to go about your usual activities without interference from your urinary problems?". Satisfact., satisfaction.
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1575 | 1593 | 1580
participants
  Baseline (BL), Any Satisfact., n=1574, 1600, 1576 | 611 | 565 | 584
  BL, Neutral /Any Dissatisfact., n=1574, 1600, 1576 | 963 | 1035 | 992
  Month (M) 12, Any Satisfact., n=1575, 1593, 1580 | 1176 | 1073 | 1114
  M12, Neutral/Any Dissatisfact., n=1575, 1593, 1580 | 399 | 520 | 466
  M24, Any Satisfact., n=1575, 1593, 1580 | 1205 | 1116 | 1088
  M24, Neutral/Any Dissatisfact., n=1575, 1593, 1580 | 370 | 477 | 492
  M36, Any Satisfact., n=1575, 1593, 1580 | 1210 | 1098 | 1074
  M36, Neutral/Any Dissatisfact., n=1575, 1593, 1580 | 365 | 495 | 506
  M48, Any Satisfact., n=1575, 1593, 1580 | 1213 | 1123 | 1043
  M48, Neutral/Any Dissatisfact., n=1575, 1593, 1580 | 362 | 470 | 537

30. Secondary Outcome: Patient Perception of Study Medication (PPSM): Number of Participants With the Indicated Responses to Question 11 (LOCF)
Description: This 12-item questionnaire (PPSM) was developed by GlaxoSmithKline for use in this study and was designed to quantify the participant's perceptions and satisfaction with the effect of study treatment on control of their urinary symptoms at baseline and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and 48. Participants were asked to respond to the question of "Overall, how satisfied are you with the study medication and it's effect on your urinary problems?". Satisfact., satisfaction.
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1574 | 1592 | 1581
participants
  Baseline (BL), Any Satisfact., n=1573, 1598, 1574 | 717 | 683 | 699
  BL, Neutral/Any Dissatisfact., n=1573, 1598, 1574 | 856 | 915 | 875
  Month (M) 12, Any Satisfact., n=1574, 1592, 1581 | 150 | 1159 | 1202
  M12, Neutral/Any Dissatisfact., n=1574, 1592, 1581 | 324 | 433 | 379
  M24, Any Satisfact., n=1574, 1592, 1581 | 1279 | 1188 | 1163
  M24, Neutral/Any Dissatisfact., n=1574, 1592, 1581 | 295 | 404 | 418
  M36, Any Satisfact., n=1574, 1592, 1581 | 1270 | 1188 | 1119
  M36, Neutral/Any Dissatisfact., n=1574, 1592, 1581 | 304 | 404 | 462
  M48, Any Satifact., n=1574, 1592, 1581 | 1262 | 1182 | 1097
  M48, Neutral/Any Dissatisfact., n=1574, 1592, 1581 | 312 | 410 | 484

31. Secondary Outcome: Patient Perception of Study Medication (PPSM): Number of Participants With the Indicated Responses to Question 12 (LOCF)
Description: This 12-item questionnaire (PPSM) was developed by GlaxoSmithKline for use in this study and was designed to quantify the participant's perceptions and satisfaction with the effect of study treatment on control of their urinary symptoms at baseline and Months 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, and 48. Participants were asked to respond to the question of "Would you ask your doctor for the medication you received in this study?".
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: as for outcome 20
Measure: Number; unit: participants
Arm/Group | Dutasteride 0.5 mg Plus Tamsulosin 0.4 mg | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Number analyzed (Participants) | 1574 | 1592 | 1581
participants
  Baseline, Yes, n=1560, 1579, 1562 | 587 | 557 | 582
  Baseline, No/Not Sure, n=1560, 1579, 1562 | 973 | 1022 | 980
  Month 12, Yes, n=1574, 1592, 1581 | 972 | 920 | 970
  Month 12, No/Not Sure, n=1574, 1592, 1581 | 602 | 671 | 611
  Month 24, Yes, n=1574, 1592, 1581 | 1027 | 955 | 952
  Month 24, No/Not Sure, n=1574, 1592, 1581 | 547 | 636 | 629
  Month 36, Yes, n=1574, 1592, 1581 | 1031 | 956 | 915
  Month 36, No/Not Sure, n=1574, 1592, 1581 | 543 | 636 | 666
  Month 48, Yes, n=1574, 1592, 1581 | 1003 | 918 | 874
  Month 48, No/Not Sure, n=1574, 1592, 1581 | 571 | 674 | 707

ADVERSE EVENTS:
Arm/Group | Combination | Dutasteride 0.5 mg | Tamsulosin 0.4 mg
Serious Adverse Events (participants affected / at risk) | 303/1610 | 339/1623 | 348/1611
Other Adverse Events (participants affected / at risk) | 618/1610 | 586/1623 | 590/1611
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination (N=1610) | Dutasteride 0.5 mg (N=1623) | Tamsulosin 0.4 mg (N=1611)
Myocardial infarction (Cardiac disorders) | 16 | 25 | 20
Coronary artery disease (Cardiac disorders) | 14 | 14 | 15
Angina pectoris (Cardiac disorders) | 14 | 14 | 15
Atrial fibrillation (Cardiac disorders) | 11 | 7 | 9
Acute myocardial infarction (Cardiac disorders) | 7 | 1 | 3
Cardiac failure (Cardiac disorders) | 5 | 1 | 5
Coronary artery stenosis (Cardiac disorders) | 4 | 5 | 2
Myocardial ischaemia (Cardiac disorders) | 3 | 3 | 3
Angina unstable (Cardiac disorders) | 1 | 3 | 4
Supraventricular tachycardia (Cardiac disorders) | 1 | 2 | 4
Acute coronary syndrome (Cardiac disorders) | 3 | 3 | 1
Bradycardia (Cardiac disorders) | 3 | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 4 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 3 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 4 | 0
Arrhythmia (Cardiac disorders) | 0 | 3 | 1
Atrial flutter (Cardiac disorders) | 1 | 1 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 1 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 1 | 0 | 1
Aortic valve disease mixed (Cardiac disorders) | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
AV dissociation (Cardiac disorders) | 0 | 1 | 0
Cardiac asthma (Cardiac disorders) | 1 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Coronary artery aneurysm (Cardiac disorders) | 1 | 0 | 0
Coronary artery thrombosis (Cardiac disorders) | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0
Cardiovascular deconditioning (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Hypertensive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Chronic left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 | 17 | 25
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 9 | 5
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6 | 4
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 5
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 3
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3
Acute myeloid leukaemia (Cardiac disorders) | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Pancreatic neolasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Retinal melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tracheal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Urinary bladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder transitional cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 11 | 15 | 8
Transient ischaemic attack (Nervous system disorders) | 5 | 5 | 4
Syncope (Nervous system disorders) | 6 | 1 | 3
Cerebral infarction (Nervous system disorders) | 1 | 4 | 3
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 4
Cerebral ischaemia (Nervous system disorders) | 3 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 2
Convulsion (Nervous system disorders) | 0 | 2 | 0
Epilepsy (Nervous system disorders) | 0 | 2 | 0
Grand mal convulsions (Nervous system disorders) | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 2 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 2 | 0
Parkinson's disease (Nervous system disorders) | 0 | 2 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 1
Brain stem ischaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Monoplegia (Nervous system disorders) | 0 | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1
Neuritis (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Senile dementia (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0 | 0
Intracranial hypotension (Nervous system disorders) | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Radicular pain (Nervous system disorders) | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral cyst (Nervous system disorders) | 0 | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 0 | 0
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 4 | 17 | 11
Abdominal pain (Gastrointestinal disorders) | 5 | 1 | 2
Colonic polyp (Gastrointestinal disorders) | 1 | 4 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal hernia (Gastrointestinal disorders) | 1 | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 2
Ileus (Gastrointestinal disorders) | 0 | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 2
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 1
Pharyngoesophageal diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Appendix disorder (Gastrointestinal disorders) | 0 | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Anal prolapse (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 13 | 10 | 6
Urniary tract infection (Infections and infestations) | 3 | 1 | 3
Cellulitis (Infections and infestations) | 3 | 3 | 0
Sepsis (Infections and infestations) | 1 | 2 | 3
Bronchitis (Infections and infestations) | 2 | 0 | 3
Diverticulitis (Infections and infestations) | 0 | 3 | 2
Lobar pneumonia (Infections and infestations) | 1 | 2 | 1
Urosepis (Infections and infestations) | 1 | 0 | 3
Bronchopneumonia (Infections and infestations) | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2
Appendicitis (Infections and infestations) | 0 | 2 | 0
Septic shock (Infections and infestations) | 0 | 2 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Device related infection (Infections and infestations) | 1 | 0 | 1
Abcess intestinal (Infections and infestations) | 0 | 1 | 0
Amoebiasis (Infections and infestations) | 0 | 1 | 0
Bronchiectasis (Infections and infestations) | 0 | 0 | 1
Carbuncle (Infections and infestations) | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 0 | 0
Epiglottitis (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0
Infective myositis (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1 | 0
Prostatic abscess (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0
Postoperative abscess (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0
Central line infection (Infections and infestations) | 0 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1
Implant site infection (Infections and infestations) | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 0
Epidemic nephropathy (Infections and infestations) | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0 | 0
Post procedural sepsis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 4 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 3 | 1 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 3 | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 2 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 3
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 2 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1 | 2
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Epicodylitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 0
Device failure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Medical device complicaiton (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural constipation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 13 | 11
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 6 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nose deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 2 | 6 | 15
Calculus ureteric (Renal and urinary disorders) | 2 | 4 | 4
Renal failure acute (Renal and urinary disorders) | 5 | 2 | 3
Calculus bladder (Renal and urinary disorders) | 0 | 3 | 4
Nephrolithiasis (Renal and urinary disorders) | 1 | 3 | 1
Renal failure (Renal and urinary disorders) | 1 | 3 | 1
Renal colic (Renal and urinary disorders) | 1 | 4 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 1
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 2
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 2
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 1 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 1
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1 | 0
Ureteral polyp (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Idioipathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Allergic granulomatous angiitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 4 | 3 | 8
Aortic aneurysm (Vascular disorders) | 3 | 2 | 1
Aortic aneurysm rupture (Vascular disorders) | 2 | 1 | 2
Aortic stenosis (Vascular disorders) | 2 | 2 | 1
Aortic dissection (Vascular disorders) | 1 | 2 | 0
Arteriosclerosis (Vascular disorders) | 1 | 2 | 0
Hypotension (Vascular disorders) | 2 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1 | 1
Peripheral ischaemia (Vascular disorders) | 2 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 1 | 0
Varicose vein (Vascular disorders) | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 2
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Malignant hypertension (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0
Venous stenosis (Vascular disorders) | 0 | 0 | 1
Arterial stenosis limb (Vascular disorders) | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Aortic dilatation (Vascular disorders) | 1 | 0 | 0
Aortic disorder (Vascular disorders) | 0 | 1 | 0
Arterial disorder (Vascular disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 4 | 6 | 6
Cholecystitis acute (Hepatobiliary disorders) | 3 | 3 | 4
Cholecystitis (Hepatobiliary disorders) | 3 | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Hydrocholecystis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 3
Non-cardiac chest pain (General disorders) | 2 | 4 | 0
Chest pain (General disorders) | 1 | 1 | 1
Multi-organ failure (General disorders) | 1 | 1 | 2
Death (General disorders) | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 1 | 0
Implant site erosion (General disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2 | 10
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 1
Epididymal cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 1
Priapism (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatic intraepithelial neoplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatism (Reproductive system and breast disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 2 | 2 | 4
Retinal detachment (Eye disorders) | 1 | 1 | 1
Macular degeneration (Eye disorders) | 1 | 0 | 2
Eye haemorrhage (Eye disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Retinal tear (Eye disorders) | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Completed suicide (Psychiatric disorders) | 1 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Chest x-ray abnormal (Investigations) | 0 | 1 | 0
Coagulation factor decreased (Investigations) | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 1 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 2 | 0 | 0
Aplasia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Hereditary sideroblastic anaemia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Purpura senile (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Arteriovenous fistula (Vascular disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination (N=1610) | Dutasteride 0.5 mg (N=1623) | Tamsulosin 0.4 mg (N=1611)
Erectile dysfunction (Reproductive system and breast disorders) | 167 | 147 | 109
Hypertension (Vascular disorders) | 133 | 147 | 136
Nasopharyngitis (Infections and infestations) | 134 | 129 | 149
Back pain (Musculoskeletal and connective tissue disorders) | 107 | 88 | 113
Influenza (Infections and infestations) | 77 | 75 | 83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.